CLINICAL TRIAL: NCT04177745
Title: The Effectiveness of Local Hot and Cold Applications on Peripheral Intravenous Catheters: A Randomised Control Trial
Brief Title: Hot and Cold Applications on PVC Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Principal İnvestigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 444
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Venous Catheterization
Keywords: Peripheral venous catheter; hot application; cold application; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hot Application (Experimental): Before PVC was inserted, the researcher applied a hot application to the catheter insertion site (inner surface of the forearm) using a hot pack for one minute. Then, the researcher made the second vein assessment and inserted a 20-G peripheral catheter into the inner surface of the forearm.
  Interventions: Other: Hot application
- Cold Application (Experimental): Before PVC was inserted, the researcher applied a cold application to the catheter insertion site (inner surface of the forearm) using a cold pack for one minute. Then, the researcher made the second vein assessment and inserted a 20-G peripheral catheter into the inner surface of the forearm.
  Interventions: Other: Cold application
- Standard Practice (No Intervention): The standard practice of the clinic was made. Accordingly, the researcher performed the vein assessment after the participants filled out the questionnaire, and then inserted the 20-G catheter into the inner surface of their forearm without any application. Afterwards, she assessed the pain and anxiety levels of the patients twice before and after the catheter insertion procedure.

INTERVENTIONS:
Other: Hot application — Before PVC was inserted, the researcher applied a hot application to the catheter insertion site (inner surface of the forearm) using a hot pack for one minute.
  Arms: Hot Application
Other: Cold application — Before PVC was inserted, the researcher applied a cold application to the catheter insertion site (inner surface of the forearm) using a cold pack for one minute.
  Arms: Cold Application

SUMMARY:
Background: This study was conducted to examine the effect of local hot and cold applications on pain, anxiety level, length of application, and vein evaluation prior to inserting PVC.

Methods: This randomised controlled trial was conducted with patients who were hospitalised in the cardiology department of a university hospital. PVC was inserted, the researcher applied a hot or cold application to the catheter insertion site for one minute.

DETAILED DESCRIPTION:
Background: This study was conducted to examine the effect of local hot and cold applications on pain, anxiety level, length of application, and vein evaluation prior to inserting PVC.

Methods: This randomised controlled trial was conducted with patients who were hospitalised in the cardiology department of a university hospital. The sample was comprised of 90 individuals, including 30 in the cold application group, 30 in the hot application group, and 30 in the control group receiving treatment in the Cardiology Clinic between November and December 2018.

ELIGIBILITY:
Inclusion Criteria:

* being able to speak and understand Turkish,
* being over 18 years of age,
* having unimpaired sense of time or place orientation,
* having no psychiatric disorders,
* having no visual or hearing problem,
* having indication of IV catheter application,
* having no administration of analgesic or anaesthetic agents prior to IV catheter insertion,
* having catheter inserted in one attempt,
* having no allergy to hot and cold applications,
* being voluntary to participate in the study.

Exclusion Criteria:

* infection
* previous history of surgery,
* scarring in the catheter insertion site,
* psoriasis in the catheter insertion site,
* active dermatitis in the catheter insertion site,
* peripheral nerve disease,
* diabetes,
* peripheral neuropathy in the catheter insertion site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale for pain and anxiety | Before catheter insertion
  The number "0" on the scale means that they do not feel any pain / anxiety and the number "10" refers to the worst pain and the highest level of anxiety.
Vein Assessment Scale | Before hot/cold application
  There are 5 assessment steps: (1) veins are neither visible nor palpable, (2) veins are visible but not palpable, (3) veins are barely visible and palpable, (4) veins are visible and palpable, and (5) veins are clearly visible and easily palpable

SECONDARY OUTCOMES:
Numeric Rating Scale for pain and anxiety | During catheter insertion
  The number "0" on the scale means that they do not feel any pain / anxiety and the number "10" refers to the worst pain and the highest level of anxiety.
Vein Assessment Scale | Immediately before insertion of the catheter
  There are 5 assessment steps: (1) veins are neither visible nor palpable, (2) veins are visible but not palpable, (3) veins are barely visible and palpable, (4) veins are visible and palpable, and (5) veins are clearly visible and easily palpable

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, Ph.D, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)